CLINICAL TRIAL: NCT00239291
Title: A Phase I/II Study of ZD1839 (Iressa) Given Concurrently With Radiotherapy in Patients With Non-Metastatic Prostate Cancer
Brief Title: Safety Study to Explore Combination of Gefitinib (ZD1839, Iressa) and Radiotherapy in Non-Metastatic Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0118
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Non-Metastatic Prostate Cancer
MeSH Terms: interventions — Gefitinib; Radiotherapy

INTERVENTIONS:
Drug: Gefitinib, radiotherapy

SUMMARY:
To estimate the safety and tolerability of 250 mg ZD1839 given concurrently with 3D-CRT in patients with non-metastatic prostate cancer

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmation of localised (T2) or locally advanced (T3) prostate cancer
* PSA below 20 ng/mL
* Lymph node negative
* Non-metastatic
* Written informed consent

Exclusion Criteria:

* Well differentiated stage T2 prostate cancer (Gleason score 2 to 4)
* Distant or nodal metastases
* Prostatectomy
* Concomitant LHRH analog treatment
* Previous or concomitant anti-androgens
* Active ILD

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2003-01; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Part A: Safety (incidence of DLTs)
Part B: Tolerability

SECONDARY OUTCOMES:
EGFR-1 expression and activation status (autophoshorylation; p-EGFR-1) at diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Finland Medical Director, MD, Study Director — AstraZeneca
Locations (1):
- Research site, Helsinki, Finland